CLINICAL TRIAL: NCT03819387
Title: A Phase I/Ib Open-Label, Multi-Center, Dose-Escalation Study to Investigate the Safety, Pharmacokinetics and Preliminary Efficacy of Intravenous NBF 006 in Patients With Non-Small Cell Lung, Pancreatic, or Colorectal Cancer Followed by a Dose Expansion Study in Patients With KRAS-Mutated Non-Small Cell Lung Cancer
Brief Title: A Study of NBF-006 in Non-Small Cell Lung, Pancreatic, or Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nitto BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBF-006-001
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Non-Small Cell Lung Cancer; Pancreatic Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NBF-006 (Experimental)
  Interventions: Drug: NBF-006

INTERVENTIONS:
Drug: NBF-006 — Intravenous infusion, once-weekly x 4 consecutive weeks, every 6 weeks

SUMMARY:
This is an open-label, non-controlled study conducted in two parts - Part A (dose escalation) followed by Part B (dose expansion).

DETAILED DESCRIPTION:
Patients in Part A will have previously treated progressive or metastatic NSCLC, pancreatic, or colorectal cancer, with or without KRAS mutation. Five dose levels will be explored. In dose level 5, only patients with previously-treated NSCLC with KRAS mutation will be included.

Patients in Part B must have previously treated NSCLC with confirmed KRAS mutation. Two dose levels will be explored further in Part B. Twenty (20) patients will be enrolled in Part B, with 10 patients enrolled in each of the two cohorts. Once dose level 5 has been confirmed to be safe in Part A (i.e. 0-1 DLT in 6 patients), an additional 4 patients will then be enrolled for a planned total of 24 patients in Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Part A: Patients with histologically or cytologically confirmed progressive or metastatic NSCLC, pancreatic, or colorectal cancer that have failed standard treatment and for which no other effective treatment is available or appropriate for the patient up to dose level 4. In dose level 5, patients with histologically or cytologically confirmed progressive or metastatic NSCLC with documented KRAS-mutant genotype, who have failed standard treatment and have no other effective treatment available or appropriate for the patient.

   Part B: Patients with histologically or cytologically confirmed progressive or metastatic NSCLC with documented KRAS-mutant genotype, who have failed standard treatment and have no other effective treatment available or appropriate for the patient.
2. Eastern Cooperative Oncology Group performance status of 0-2.
3. Men and women ≥ 18 years of age.
4. Patients must have recovered from all acute adverse effects (excluding alopecia) of prior therapies to baseline or ≤ Grade 1 prior to study entry.
5. Adequate bone marrow function, defined as an absolute neutrophil count (ANC) ≥ 1.5 x 109/L and a platelet count ≥ 100 x 109/L.
6. Adequate renal function, defined as serum creatinine ≤ 1.5 x upper limit of normal (ULN) for the institution or calculated creatinine clearance [Cockcroft-Gault method] must be ≥ 60 mL/min/1.73 m². If serum creatinine is >1.5 x ULN, then creatinine clearance can be calculated from a 24-hour urine collection.
7. Adequate hepatic function, defined as total bilirubin ≤ 1.5 mg/dL and alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 x ULN, or ≤ 5 x ULN if known liver metastases.
8. Female patients of childbearing potential must have a negative serum or urine pregnancy test result at time of pre-treatment screening.
9. Patients with reproductive potential must agree to use at least one form of highly effective contraception prior to study entry and for up to 30 days beyond the last administration of study drug.
10. Patients must be capable of providing informed consent and must be willing to provide written informed consent prior to the start of any study-specific procedures.
11. All patients must have measurable tumor per RECIST 1.1.
12. Agree to adhere to all study protocol requirements.

Exclusion Criteria:

1. Prior chemotherapy, radiation therapy, or investigational therapy within 4 weeks (exception: 6 weeks for nitrosoureas or mitomycin C); or prior non-cytotoxic therapy within 5 drug half-lives (or 4 weeks, whichever is shorter); or monoclonal antibodies within 4 weeks prior to the first dose of study treatment.
2. Concurrent use of any other investigational agent.
3. Known or clinically suspected central nervous system or leptomeningeal metastases, unless irradiated or treated a minimum of 4 weeks prior to first study treatment and stable without requirement of corticosteroids for > 1 week.
4. Pregnant or breast feeding. A negative pregnancy test must be documented at baseline for women of childbearing potential. Patients may not breast-feed infants while on this study.
5. Significant cardiovascular disease or condition, including:

   1. Congestive heart failure currently requiring therapy
   2. Need for antiarrhythmic medical therapy for ventricular arrhythmia
   3. Severe conduction disturbance
   4. Angina pectoris requiring therapy
   5. QTc interval > 450 msec (males) or > 470 msec (females) Fridericia's correction.

      Note: QTc values up to 500 ms will be acceptable where patient's medical history e.g. bundle branch block, is known to cause mild QTc prolongation and the condition is well controlled.
   6. History of congenital long QT syndrome or congenital short QT syndrome
   7. Uncontrolled hypertension (per the Investigator's discretion)
   8. Class III or IV cardiovascular disease according to the New York Heart Association's Functional Criteria
   9. Myocardial infarction within 6 months prior to first study drug administration
6. Known history of human immunodeficiency virus or active infection with hepatitis B virus or hepatitis C virus.
7. Known uncontrolled intercurrent illnesses, including uncontrolled viral influenza and COVID 19, systemic bacterial infections, and fungal infections.
8. Psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies.
9. Known allergic reactions to H1/H2 antagonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by CTCAE v5.0 | Change in the incidence and severity of adverse events related to study treatment from baseline to 4 weeks following last dose

SECONDARY OUTCOMES:
Best Overall Response per RECIST 1.1 | Number of days from date of first dose to 30 days after last treatment
  The rate of complete remission (CR) + partial remission (PR) + stable disease (SD)
Pharmacokinetic parameters for siRNA | Up to 72 hours from start of infusion on Cycle 1, Day 1 and Day 22 and prior to infusion Cycle 1, Day 8 and Cycle 2, Day 1
  Peak Plasma Concentration (Cmax)
Additional pharmacokinetic parameters for siRNA | Up to 72 hours from start of infusion on Cycle 1, Day 1 and Day 22 and prior to infusion Cycle 1, Day 8 and Cycle 2, Day 1
  Area under the plasma concentration versus time curve (AUC)

OTHER OUTCOMES:
To evaluate correlation between biomarkers and clinical outcome | Number of days from date of first dose to 30 days after last treatment
  analysis of ADAs, immune activation biomarkers, GSTP knockdown, and other biomarker activity
To evaluate correlation between KRAS mutations and clinical outcome | Number of days from date of first dose to 30 days after last treatment

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Toledo, Eleanor N. Dana Cancer Center, Toledo, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - NEXT Oncology - Austin, Austin, Texas
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - NEXT Oncology - San Antonio, San Antonio, Texas
  - NEXT Oncology - Virginia, Fairfax, Virginia

DOCUMENTS (3):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03819387/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT03819387/SAP_001.pdf
  • Informed Consent Form (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT03819387/ICF_002.pdf